CLINICAL TRIAL: NCT06294457
Title: Effectiveness of Non-invasive Neuromodulation Treatment (NESA) for the Management of Constipation Without Diagnosed Pathology in Students of the European University of Madrid (Spain)
Brief Title: Effectiveness of Non-invasive Neuromodulation for Intestinal Transit in Healthy Subjects
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Europea de Madrid (Other)
Responsible Party: Principal Investigator, Vanesa Abuín, Associated Professor, Universidad Europea de Madrid
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: CI-2024-480
Record Dates: First submitted 2024-02-19; First posted 2024-03-05 (Actual); Last update posted 2024-03-05 (Actual); Status verified 2024-03

CONDITIONS: Constipation
MeSH Terms: conditions — Constipation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: The device will be placed with no current. This type of neuromodulation gives no feeling at all to the patient while administred, so there is no way for the patient to know if the apparatus is connected or not.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): The total number of sessions to be conducted for each patient will be 10 sessions, spread over 5 weeks, which means a frequency of twice a week.
  Each NESA microcurrent session will last 60 minutes. A maximum time of 15 minutes will be allowed for connecting the patient at the beginning and for removing the device at the end.
  The directing electrode will be located throughout the treatment between the spinous processes of C6 and C7 to act generally on the individual, and in later sessions, the electrode will be placed d at T12-S3 to influence the sacral plexus.
  The intensity will be set to Low (3 volts) in all sessions,. The other device parameters range between 100-900 microamperes and between 1.14 and 14.29 hertz, and are preset by each program.
  Interventions: Device: Non-Invasive Neuromodulation NESA
- Placebo (Placebo Comparator): Non-active Non-Invasive Neuromodulation NESA
  Interventions: Device: Non-Invasive Neuromodulation NESA

INTERVENTIONS:
Device: Non-Invasive Neuromodulation NESA — Considering the objectives set: In the first phase, the directing electrode will be located at C6-C7 to generate a systemic and general effect on the organism, with program 1, program 2, program 7, and program 8. In the second phase, the directing electrode will be placed at the abdominal level in the area of the mesenteric plexus to influence the sympathetic innervation of the viscera. In the third phase, the directing electrode is located at S2-S3 to concentrate the action of the therapy on the sacral parasympathetic plexus, responsible for the innervation of the rectum. In this way, both the sympathetic and parasympathetic innervation of the main sexual organs and the large intestine are covered through the sympathetic paravertebral ganglia and the sacral plexus.

SUMMARY:
Objectives

Main objective:

Assess the effectiveness of non-invasive neuromodulation treatment (NESA) for the management of constipation in patients without diagnosed pathology in Spain

Secondary objectives:

Evaluate the improvement in sleep quality Analyze the improvement in blood pressure quality Measure the improvement in cortisol quality Determine if there is an improvement in heart rate

DETAILED DESCRIPTION:
Background and Current State of the Topic Non-invasive NESA neuromodulation is based on a superficial treatment through electrical microcurrents, regulated by Wilder's law and hormesis.

It involves applying a low-frequency biphasic current that emits up to 19,000 pulses/minute, with an intensity varying from 0.1 to 1 milliwatt and a frequency from 1 to 15 hertz, generating a weak and physiological electrical signal which is amplified due to its entry through many pathways via electrodes placed on the limbs .

Imperceptible sensations are produced in areas of low impedance for individuals. All these parameters fluctuate according to the device's programs. NESA aims to neuromodulate the Autonomic Nervous System (ANS), inducing changes in the endogenous responses of dysfunctional systems or those with pathologies. The ANS is an essential component of the Nervous System responsible for maintaining the organism's homeostasis and responding to internal or external changes through adaptation responses. It consists of the sympathetic and parasympathetic systems, involuntary systems in charge of regulating respiration, circulation, metabolism, digestion, body temperature, reproduction, and glandular secretion.

Constipation is defined as a gastrointestinal motility disorder characterized by difficult or infrequent bowel movements (fewer than three times per week). It is one of the most common gastrointestinal diseases, affecting between 0.7% and 29.6% of the population in developed and developing countries. Constipation can affect overall quality of life. It may trigger sleep disorders, anxiety, depression, and other psychological complications, even increasing mortality associated with conditions such as hypertension, cardiovascular diseases, cerebrovascular diseases, and the incidence of colon cancer.

Since the etiology and mechanism of constipation are complicated, many of the currently available treatments are not effective for many people.

Given that NESA performs a non-invasive neuromodulation on the ANS through the nerve pathways involved in improving constipation, effects in this regard are expected.

Non-invasive NESA neuromodulation has emerged as a promising area of research with potentially significant results in terms of improving sleep quality and daytime sleepiness, nerve and cognitive function, quality of life, and pain. This study aims to clarify these aspects, establishing a solid foundation for clinical practice and future research.

Justification The ANS is responsible for maintaining the organism's homeostasis and responding to internal or external changes through adaptation responses. The gastrointestinal motility disorder of constipation and the irregular contractions of overactive bladder are conditions in which there are alterations in the ANS, which is why neuromodulation of the ANS can induce changes in the endogenous responses in dysfunctional systems . The chosen population is healthy or not previously diagnosed to assess them for changes in gastrointestinal motility

ELIGIBILITY:
Inclusion Criteria:

* Participants from 18 to 65 years old
* Sign informed consent

Exclusion Criteria:

* Diagnosed diseases at the time of the study.
* Severe previous psychiatric conditions.
* Medical contraindications that prevent the use of non-invasive neuromodulation therapy.
* Having exercised in the hours prior to the NESA treatment.
* Having consumed coffee or tobacco in the hours prior to the treatment.
* Minors.
* Individuals who have previously received any type of neuromodulation treatment.
* Cancer.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-03 (Estimated); Primary Completion 2024-03 (Estimated); Study Completion 2024-06 (Estimated)

PRIMARY OUTCOMES:
Quality of life by constipation (CVE-20) | 10 minutes
  Questionnaire. https://www.sciencedirect.com/science/article/abs/pii/S0025775308722851#aep-article-footnote-id

SECONDARY OUTCOMES:
Sleep Quality | 10 minutes
  Questionnaire
Cardiac Frecuency | 5 minutes
  Measured with WeCardio.
Arterial pressure | 5 minutes
  With Sfigmomanometer

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Citation — https://www.frontiersin.org/articles/10.3389/fphys.2022.1032020
- See also: Citation — https://www.cientperiodique.com/article/CPQOS/5/4/97
- See also: Citation — https://doi.org/10.1016/j.eurpsy.2016.01.578
- See also: Citation — https://doi.org/10.1016/j.eurpsy.2017.01.1048
- See also: Citation — https://doi.org/10.1186/s12887-023-04307-4